CLINICAL TRIAL: NCT05860634
Title: Urinary Catheter Self-Discontinuation After Urogynecology Surgery
Acronym: CATH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004321
Record Dates: First submitted 2023-04-27; First posted 2023-05-16 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-01

CONDITIONS: Urinary Retention; Pelvic Organ Prolapse; Stress Urinary Incontinence; Catheter Related Complication
Keywords: Post-operative urinary retention; Pelvic organ prolapse; Stress urinary incontinence; Cather self-discontinuation
MeSH Terms: conditions — Urinary Retention; Pelvic Organ Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Catheter office-discontinuation group (No Intervention): The patients randomized to the office-discontinuation group will visit the office for a repeat voiding trial on postoperative day 1. At this visit, the patients will undergo a backfill voiding trial.
- Catheter self-discontinuation group (Experimental): The patients randomized to the catheter self-discontinuation group will be provided with a diagrammatic handout and will be instructed to remove their indwelling urinary catheter at home on the morning of Postoperative day 1.
  Interventions: Procedure: Catheter self-discontinuation

INTERVENTIONS:
Procedure: Catheter self-discontinuation — Self-discontinuation of a transurethral catheter
  Arms: Catheter self-discontinuation group

SUMMARY:
The goal of this randomized clinical trial is to determine if removal of transurethral urinary catheters by patients at home is as safe as catheter removal in the office following urogynecologic surgery.

Participants will be randomized to either standard catheter removal in the office or catheter self-removal at home.

DETAILED DESCRIPTION:
This is a prospective, randomized, two-parallel arm, non-inferiority trial to evaluate two methods of catheter discontinuation in women with post-operative urinary retention (POUR) after surgery for pelvic organ prolapse (POP) or stress urinary incontinence (SUI). This study will evaluate whether self-discontinuation of transurethral catheter by patients is non-inferior to standard office discontinuation based on rates of persistent POUR on post-operative day (POD) 1.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years of age
2. Are fluent and able to read in English or Spanish
3. Undergo POP and/or SUI surgery (uterosacral ligament suspension, sacrospinous ligament fixation, sacral colpopexy, anterior colporrhaphy, posterior colporrhaphy, and/or mid-urethral sling) that occurs on Monday - Thursday
4. Have transurethral catheter in place at the conclusion of surgery as part of standard care
5. Are diagnosed with POUR on POD0 based on ultrasound bladder scan PVR of 100 mL or more
6. Are discharged home on the same day of surgery (POD 0)

Exclusion Criteria:

1. Have preoperative voiding dysfunction requiring self-catheterization or indwelling transurethral catheter
2. Have physical or mental impairment that would impact their ability to remove their catheter themselves.
3. Undergo urethral bulking injections as part of surgery
4. Have undergone a planned or unplanned urinary tract procedure requiring prolonged catheterization as standard of care (e.g. cystotomy repair, ureteral reimplantation, vesicovaginal fistula repair, urethral diverticulum repair)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Postoperative Urinary Retention | Post-operative day 1
  Non-inferiority comparison of the rates of persistent POUR on POD1 between catheter self-discontinuation and standard office catheter. Persistent POUR is defined as PVR greater than 100 mL by bladder scan on POD1.

SECONDARY OUTCOMES:
Rates of postoperative urinary tract infection (UTI) | within 6 weeks of surgery
  Rates of postoperative UTI within 6 weeks of surgery - UTI will be defined as treatment with antibiotics for symptoms of UTI.
Incidence of recurrent POUR | within 6 weeks of surgery
  Recurrent POUR will be defined as any participant with successful POD1 voiding trial who later requires replacement of catheter due to recurrent POUR within 6 weeks of surgery. Recurrent POUR is defined as PVR greater than 100 mL by bladder scan after passing initial POD1 voiding trial.
Number of postoperative patient encounters | within 6 weeks of surgery
  Number of postoperative patient encounters, including any patient call to the office, electronic medical record message to office from patient, office visit, or emergency department visit.
Patient satisfaction assessment via the Acceptability of Intervention Measure (AIM) Questionnaire | Post-operative day 1
  Patient satisfaction with catheter removal method as assessed via the Acceptability of Intervention Measure (AIM) Questionnaire.
  The AIM Questionnaire is a 4-item questionnaire on a 5-point Likert scale. Response Scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree Scoring Instructions: Scale is created by averaging responses. Scale values range from 1 to 5.
  The higher the score is, the higher the degree the patient finds the intervention acceptable.
Patient satisfaction assessment via the the Surgical Satisfaction Questionnaire - 8 (SSQ-8). | Post-operative day 1
  Patient satisfaction with catheter removal method as assessed via the Surgical Satisfaction Questionnaire - 8 (SSQ-8).
  The SSQ-8 is an 8-item questionnaire, with responses recorded on a 5-point Likert scale with responses from 0 "Very Unsatisfied" to 4 "Very Satisfied." Scoring uses the mean average of the 8 scores being multiplied by 25 (the questionnaire is considered incomplete if more than 2 items are not answered), yielding a potential range of scores from 0 to 100. The higher the score is, the greater the degree of surgical satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Rieger, MD, Principal Investigator — University of Texas at Austin; Collin M McKenzie, MD, Principal Investigator — University of Texas at Austin
Locations (4):
- United States (4):
  - University of Texas of Austin - Dell Seton Medical Center, Austin, Texas
  - Seton Medical Center Austin, Austin, Texas
  - Ascension Seton Hays Hospital, Kyle, Texas
  - Seton Medical Center Williamson, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: No